CLINICAL TRIAL: NCT04203745
Title: Clinical Evaluation of a Nonablative Fractional 1940 nm Diode Laser for Skin Resurfacing and Treatment of Pigmented Lesions
Brief Title: Nonablative Fractional Diode Laser for Treatment of Skin Resurfacing and Pigmented Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Candela Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FRX19004
Record Dates: First submitted 2019-12-10; First posted 2019-12-18 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Skin Texture; Pigmented Lesions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Nonablative Fractional Diode Laser (Experimental): Single Group - single arm study. Group was treated with Nonablative Fractional Diode Laser
  Interventions: Device: Nonablative Fractional Diode Laser

INTERVENTIONS:
Device: Nonablative Fractional Diode Laser — The FRAX 1940 is a fractional 1940 nm solid-state diode laser that delivers linear arrays of microbeams to create nonablative microscopic treatment zones (MTZs) in the skin.

SUMMARY:
This study is intended to evaluate the efficacy and safety of a new diode fractional laser for skin resurfacing and treatment of pigmented lesions.

DETAILED DESCRIPTION:
This study is a prospective, open-label, clinical trial to study the effects of the nonablative, fractional diode laser for skin resurfacing.

Up to 60 eligible participants will be enrolled at up to three (3) sites. Participants will receive up to 4 treatments to the face, and other off-face locations may be treated. Participants will complete follow-up visits for clinical evaluation and photography at 1 and 3 months after the final treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female
2. Age 21 to 70
3. Fitzpatrick Skin Type I to V
4. Willingness to have test spots and up to three (3) skin resurfacing treatments on the face
5. Presence of pigmented lesions to be treated off the face must be rated at baseline as moderate or higher per Investigator or study staff
6. Provide signed informed consent to participate in the study
7. Adhere to study treatment and follow-up schedules
8. Willing to have hair removed from the intended treatment area prior to treatment and/or photography
9. Avoid sun exposure to all treated areas and use of sunscreen with sun protection factor (SPF) 30 or greater throughout the duration of the study
10. Adhere to post-treatment care instructions
11. Allow photography of treated areas and to release their use for scientific and/or promotional purposes

Exclusion Criteria:

1. Pregnant, planning to become pregnant, or breast feeding during the study
2. Allergy to lidocaine or similar medications
3. Excessively tanned skin in the intended treatment area
4. Open wound or infection in the intended treatment area
5. Tattoo(s) or permanent make-up in the intended treatment area
6. Skin condition in the intended treatment area that could interfere with treatment or evaluation of safety or efficacy
7. Presence or history of melasma
8. Presence or history of skin cancer within the treatment area(s)
9. History of keloid or hypertrophic scar formation
10. History of herpes simplex virus (HSV) or similar condition in the intended treatment area unless treated with prophylactic medication
11. Diagnosed coagulation disorder
12. Immunosuppression
13. Presence of any medical condition that in the opinion of the Investigator could impair healing or outcome as a result of treatment
14. Use of systemic retinoid therapy (e.g. Accutane) during the past six (6) months
15. Use of topical retinoid therapy in the intended treatment area during the past two (2) weeks
16. Use of oral corticosteroid therapy during the past four (4) weeks
17. Prior skin resurfacing treatment, such as surgery, light, laser or radiofrequency (RF) procedures in the intended treatment area during the past six (6) months
18. Prior injectable dermal fillers in the intended treatment areas within the past twelve (12) months
19. Prior injectable toxins (Botox) in the treated areas within the past three (3) months
20. Subjects who in the opinion of the Investigator are unwilling or unable to adhere to the study requirements, or who are otherwise not a good candidate for the study

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Konika P Schallen, M.D., Principal Investigator — Candela Corporation
Locations (1):
- Candela Institute for Excellence, Marlborough, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Nonablative Fractional Diode Laser: Single Group - single arm study
  Nonablative Fractional Diode Laser: The FRAX 1940 is a fractional 1940 nm solid-state diode laser that delivers linear arrays of microbeams to create nonablative microscopic treatment zones (MTZs) in the skin.
Period: Overall Study
Arm/Group | Nonablative Fractional Diode Laser
Started | 26
Completed | 20
Not Completed | 6

BASELINE CHARACTERISTICS:
Population: 26 subjects with 36 areas were enrolled in study FRX19004
Units Other Than Participants: treatment areas
Groups:
- Single Group: Single Group - single arm study
  Nonablative Fractional Diode Laser: The FRAX 1940 is a fractional 1940 nm solid-state diode laser that delivers linear arrays of microbeams to create nonablative microscopic treatment zones (MTZs) in the skin.
Arm/Group | Single Group
Number analyzed (Participants) | 26
Number analyzed (treatment areas) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 11
  Caucasian (White) | 15
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Pigmented Lesion Improvement by Blinded Evaluation
Description: The primary efficacy endpoint was defined as improvement in the clearance of pigmented lesions, as assessed by three (3) blinded evaluators comparing photographs taken at Baseline/Pre-treatment and at the 1-month follow-up (post final treatment)
Time Frame: 1 month follow-up post treatment series, where treatment could last up to 10 weeks from baseline
Population: Data from FRX19004 study was combined with FRX19005 study (NCT04202419) for ad-hoc primary efficacy analysis via blinded evaluation. Both trials assessed the 'treatment of pigmented lesions' and are directly comparable due to equivalence of patient populations and efficacy endpoints, therefore, the exact same analyses were performed. The treated area was considered a "success" if at least 2 of the 3 reviewers correctly identified the post-treatment photograph (i.e. left or right side).
Measure: Count of Units; unit: observations
Units Other Than Participants: observations
Arm/Group | Nonablative Fractional Diode Laser
Number analyzed (Participants) | 56
Number analyzed (observations) | 45
observations | 41

ADVERSE EVENTS:
Time Frame: 12 weeks following last treatment, where treatment series could last up to 10 weeks.
Arm/Group | Single Group
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 4/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Group (N=26)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Melasma (Skin and subcutaneous tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-30): https://cdn.clinicaltrials.gov/large-docs/45/NCT04203745/Prot_SAP_001.pdf